CLINICAL TRIAL: NCT04782713
Title: Smart PSA Screening Study
Brief Title: Smart Prostate Specific Antigen (PSA) Screening Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Peter Gann, Principal Investigator, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2020-1251
Record Dates: First submitted 2021-02-03; First posted 2021-03-04 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: PSA; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a single-arm intervention with historical control trial where the direct recipients of the intervention are PCPs. There are three components to the project with corresponding data collection activities - I) PCP Evaluation of the Smart PSA Screening Guidelines
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PCP Evaluation of Smart PSA Screening Guidelines (Other): Completing surveys at baseline, 3, 6, 9 and 12 months
  Interventions: Other: Completing surveys

INTERVENTIONS:
Other: Completing surveys — Completing surveys at baseline, 3, 6, 9, and 12 months

SUMMARY:
This intervention includes the introduction of the Prostate Cancer Working Group (PCWG )Smart PSA Screening Guidelines and implementation of patient navigation/ care coordination for men with elevated PSA (>4.0 ng/mL).

The guidelines include:

1. What age to start?
2. How often to repeat screening?
3. What age to stop?
4. What PSA threshold should trigger a biopsy referral?

DETAILED DESCRIPTION:
Primary care providers (PCP) hold the key to implementing effective early detection of Prostate Cancer (PCa), but uncertainty about how to use PSA for screening without causing undue overtreatment of indolent cancer, has greatly inhibited implementation, even in high-risk communities. This is a single-arm intervention study to test implementation of the Smart PSA strategy plus system-level patient navigation/ care coordination in the Mile Square Health Center(MSHC), in order to: a) identify barriers and facilitators to inform implementation of care, b) evaluate the impact on provider confidence regarding prostate cancer screening, and, c) measure its effect on observed PSA levels, biopsy referral rates, and biopsy outcomes.

100 PCPs employed by MSHC who provide care for male adults will be asked to participate in surveys at baseline, (prior to an in-service training) and at 3,6, 9 and 12 months. The surveys will use 5-point Likert scales to assess the respondent's self-report of their knowledge regarding PSA screening, attitudes, behavior; and confidence in presenting the issue, discussing it with patients, interpreting results and making recommendations based on them; and to elicit comments on how to improve implementation.

Historical data of 4500 patients covering a one year period prior to the intervention will be used to measure the impact of the intervention on measurable outcomes

ELIGIBILITY:
Inclusion Criteria for PCP:

* PCP employed by MSHC who provides care for male adult patients

Exclusion Criteria for PCP:

* Not a PCP employed by MSHC who provides care for male adult patients

Inclusion Criteria for Patient navigator/care coordinator:

* Male
* Age 40-75
* Clinic visit at a MSHC site
* Elevated PSA (>4.0 ng/ml)

Exclusion Criteria for Patient navigator/care coordinator:

• Not meeting the inclusion criteria

Inclusion criteria for chart and database review:

* Male
* Age 40-75
* Clinic visit at a MSHC site from date of study start through 12 months (comparison of 12-month intervention period to periods before and after intervention implementation)

Exclusion Criteria for chart and database review:

• Not meeting the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Number of PSA tests ordered per number of clinical encounters 12 months prior to the intervention | Monthly for 12 months prior to intervention
  Review Pathology Laboratory Services, Ambulatory Services Administration, UI Health for PSA orders
Number of PSA tests ordered per number of clinical encounters during the intervention | Monthly for 12 months during intervention
  Review Pathology Laboratory Services, Ambulatory Services Administration, UI Health for PSA orders
Number of PSA levels categorized as <4.0, 4.0-10.0 and >10.0 12 month prior to the intervention | Monthly for 12 months prior to intervention
  Review Pathology Laboratory Services, UI Health PSA results
PSA levels categorized as <4.0, 4.0-10.0 and >10.0 during the intervention | Monthly for 12 months during intervention
  Review Pathology Laboratory Services, UI Health PSA results
Number of Urology referrals 12 months prior to the intervention | 12 months prior to intervention
  Review electronic medical records for urology referrals
Number of Urology referrals during the intervention | 12 months after intervention
  Review electronic medical records for urology referrals
Number of prostate biopsies performed using the risk levels of the National Comprehensive Cancer Network (NCCN) of very low, Favorable intermittent, Unfavorable intermittent, High, very high 12 months prior to the intervention | 12 months prior to the intervention
  Review electronic medical records for biopsies performed
Number of prostate biopsies performed using the risk levels of the National Comprehensive Cancer Network (NCCN) of very low, Favorable intermittent, Unfavorable intermittent, High, very high during the intervention | 12 months after the intervention
  Review electronic medical records for biopsies performed
Number of prostate biopsy complications 12 months prior to the intervention | 12 months prior to intervention
  Review electronic medical records and pharmacy database for biopsy complications using NCI Common Toxicity Criteria to rate complications from mild to life-threatening
Number of prostate biopsy complications during the intervention | 12 months after intervention
  Review electronic medical records and pharmacy database for biopsy complications using NCI Common Toxicity Criteria to rate complications from mild to life-threatening
Benefit and harm analysis 12 months prior to the intervention | 12 months prior to intervention
  Assess the Cancer of the Prostate Risk Assessment (CAPRA) score and National Comprehensive Cancer Network (NCCN) risk levels for each patient diagnosed per NCCN: Very Low, Low, Favorable intermediate, Unfavorable Intermediate, High, Very High. Subgroup analyses by age, race and previous screening history will be performed. Attention will be focused on relative changes in the number of clinically significant but treatable cases to the number of clinically insignificant cases. Clinically significant but treatable cases will be defined as NCCN Intermediate (thus all localized Gleason 7); clinically insignificant cases will be defined as NCCN Very Low (PSA<10, Gleason grade ≤ 6, T1c, < 3 positive cores, no core > 50% cancer, PSA density < 0.15
Benefit and harm analysis 12 months prior to the intervention | 12 months prior to intervention
  Assess the Cancer of the Prostate Risk Assessment (CAPRA) score and National Comprehensive Cancer Network (NCCN) risk levels for each patient based on age and race
Benefit and harm analysis 12 months prior to the intervention | 12 months prior to intervention
  Assess the Cancer of the Prostate Risk Assessment (CAPRA) score and National Comprehensive Cancer Network (NCCN) risk levels for each patient based on previous screening history
Benefit and harm analysis 12 months prior to the intervention | 12 months prior to intervention
  Compare the number of clinically significant but treatable cases to the number of clinically insignificant cases. Clinically significant but treatable cases will be defined as NCCN Intermediate with localized Gleason grade 7, clinically insignificant cases will be defined as NCCN Very Low PSA<10, Gleason grade ≤ 6, T1c, < 3 positive cores, no core > 50% cancer, PSA density < 0.15
Benefit and harm analysis during the intervention | 12 months after intervention
  Assess the Cancer of the Prostate Risk Assessment (CAPRA) score and National Comprehensive Cancer Network (NCCN) risk levels for each patient diagnosed per NCCN: Very Low, Low, Favorable intermediate, Unfavorable Intermediate, High, Very High.
Benefit and harm analysis during the intervention | 12 months after intervention
  Assess the Cancer of the Prostate Risk Assessment (CAPRA) score and National Comprehensive Cancer Network (NCCN) risk levels for each patient based on age and race
Benefit and harm analysis during the intervention | 12 months after intervention
  Assess the Cancer of the Prostate Risk Assessment (CAPRA) score and National Comprehensive Cancer Network (NCCN) risk levels for each patient based on previous screening history
Benefit and harm analysis during the intervention | 12 months after intervention
  Compare the number of clinically significant but treatable cases to the number of clinically insignificant cases. Clinically significant but treatable cases will be defined as NCCN Intermediate with localized Gleason grade 7, clinically insignificant cases will be defined as NCCN Very Low PSA<10, Gleason grade ≤ 6, T1c, < 3 positive cores, no core > 50% cancer, PSA density < 0.15
Number of PCPs that have confidence in discussing prostate issues 12 months prior to the intervention | 12 months prior to intervention
  Analyses of graphing mean trajectories in response to repeat surveys among PCPs at baseline, 3, 6, 9 and 12 months. Subgroup analyses will compare responses stratified by gender, years in practice, race and site
Number of PCPs that have confidence in discussing prostate issues during the the intervention | 12 months after intervention
  Analyses of graphing mean trajectories in response to repeat surveys among PCPs at baseline, 3, 6, 9 and 12 months. Subgroup analyses will compare responses stratified by gender, years in practice, race and site
Number of patients referred to specialty care 12 months prior to patient navigation/ care coordination | 12 months prior to intervention
  Review electronic medical records for referral to specialty care
Number of patients referred to specialty care through patient navigation/ care coordination during the intervention | 12 months after intervention
  Review electronic medical records for referral to specialty care

CONTACTS AND LOCATIONS:
Overall Officials: Peter Gann, MD, ScD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- Mile Square Health Center, Chicago, Illinois, United States